CLINICAL TRIAL: NCT03576534
Title: Pre Bypass Ultrafiltration (PBUF) Improves Intraoperative Glucose, Sodium, Potassium and Lactate Levels in Children Requiring Cardiopulmonary Bypass
Brief Title: Pre Bypass Ultrafiltration (PBUF) in Children Requiring Cardiopulmonary Bypass
Acronym: PBUF
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Given SARS CoV2 pandemic, we had difficulty enrolling patients in the proposed time frame
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Meena Nathan, Staff Surgeon, Department of Cardiac Surgery, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P00028603
Record Dates: First submitted 2018-05-29; First posted 2018-07-03 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Congenital Heart Disease
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Intervention Model Description: Randomized Control Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Standard of care
- Study (Active Comparator): PBUF used prior to Cardiopulmonary bypass
  Interventions: Other: Use of prebypass ultrafiltration (PBUF)

INTERVENTIONS:
Other: Use of prebypass ultrafiltration (PBUF) — In addition to standard of care for cardiopulmonary bypass, in the study arm prebypass ultrafiltration will be performed.
  Arms: Study

SUMMARY:
Newborn babies and children with congenital heart defects who need heart surgery need to be placed on the heart-lung machine for heart surgery.

In order to use the heart-lung machine, the investigators have to use blood and other fluids to fill the tubing. During the operation, ultrafiltration is carried out as standard of care to remove extra fluid. Modified ultrafiltration is also performed after surgery. In this study, the investigators are looking to use the filter additionally before surgery. Using the pre bypass filtration before the subject is placed on the heart-lung machine will allow the investigators to better normalize electrolytes in the blood/fluid mixture used in the heart lung machine. This technique is called pre-bypass ultrafiltration, or PBUF (pronounced "P" Buff).

The investigators are conducting a study to see if using PBUF to better normalize electrolytes in the blood will make a difference. The investigators have been adding fluids to prime the heart-lung machine in two different ways. The investigators believe both methods are safe and acceptable but hypothesize that there may be subtle differences in electrolytes and fluid status when one technique is used as opposed to the other. The investigators believe that neither technique introduces risk since both are currently used in practice. The standard method adds blood to the heart-lung machine. The alternate method adds blood to the heart-lung machine and then additional fluid is added and removed to more normalize the electrolytes. The investigators plan to randomized subjects undergoing heart surgery to receive the standard priming method versus PBUF to determine if there is any difference in outcomes. Laboratory and clinical data collected as part of clinical care will be used to determine difference sin outcomes. There will be no additional blood taken for this study.

There are no known risks to PBUF. The benefits include helping investigators determine if PBUF does or does not make a difference to how subjects recover after surgery. The investigators believe that providing more normal blood values will either improve the subjects' outcome or have no benefit. The investigators do not anticipate increased risks.

Given COVID -19 restrictions, the study is on hold.

DETAILED DESCRIPTION:
Research question: Can PBUF provide more physiologic values for glucose, sodium, potassium and lactate throughout the cardiopulmonary bypass period without an increased incidence of adverse events?

Background: The values for glucose, sodium, potassium and lactate in blood primes for subjects weighing less than 8 kg are known to be non-physiologic. The process of priming the cardiopulmonary bypass circuit is not standardized across institutions and there are several methods used to correct for known prime value issues. The investigators documented the prime values for 20 subjects weighing less than 8 kg and then performed pre-bypass ultrafiltration (PBUF) on the prime for those same circuits to achieve more physiologic prime values. The investigators were cautious not to implement too significant of a change as the investigators assessed the technique and documented that plasma-free hemoglobin importantly did not rise and that measured osmolality was still slightly above the normal range.

Study type: Prospective randomized controlled study.

Hypothesis: The investigators hypothesize that pre cardiopulmonary bypass ultrafiltration (PBUF) can provide more physiologic prime values for glucose, sodium, potassium and lactate. Plasma-free hemoglobin will not increase with the technique. Osmolality will be maintained slightly above the normal range. PBUF will not negatively impact clinical outcome measures and may improve them.

Specific Aim 1 To determine if use of PBUF will result in more physiologic values for glucose, sodium, potassium and lactate during and immediately after cardiopulmonary bypass.

Specific Aim 2 To determine if PBUF can be achieved with no increase in plasma free hemoglobin while maintaining plasma osmolality within acceptable range during and immediately after cardiopulmonary bypass.

Specific Aim 3 To determine if use of PBUF will result in improved clinical outcomes after surgery on cardiopulmonary bypass.

Randomization: Prior to surgery, subjects will be randomized to one of the two study groups using a randomly permuted blocks design.

Statistical analysis: Analyses will be performed on an intention to treat basis. Comparisons of subject characteristics and outcomes will be made using the two-sample t test or Wilcoxon rank sum test for continuous variables, and Fisher's exact test for categorical variables. If imbalances in patient factors exist between the two groups, linear and logistic regression will be used to compare outcomes for the groups adjusting for these potential confounders.

Sample size calculation: Sample size is calculated for comparisons of subjects in the normal range of values for the PBUF and standard care groups. This will be done separately for glucose, sodium, potassium, and lactate; each comparison will be performed at the 0.0125 level of significance. If 70% of standard care subjects are in the normal range versus 90% of PBUF subjects, a total of 176 subjects (88 per group) would be required to achieve 80% power. With 350 eligible subjects that meet inclusion criteria based on 2017 numbers and 75% consent rate the investigators will be able to enroll 260 subjects in 1 year.

Given COVID-19 restrictions, the study is on hold.

ELIGIBILITY:
Inclusion Criteria:

* All patients < 8 kilograms and < 1 year (to ensure that all patients receive steroids at initiation of CPB) undergoing an index cardiac operation for that hospitalization (using a single PBUF protocol)

Exclusion Criteria:

* Patients undergoing repeat cardiac surgery within the same admission
* Patients undergoing transplants as their index surgery
* Patients undergoing Ventricular assist device implantation as their index surgery

Ages: 1 Day to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 13 (Actual)
Dates: Start 2019-10-03 (Actual); Primary Completion 2021-09-13 (Actual); Study Completion 2021-09-13 (Actual)

PRIMARY OUTCOMES:
Glucose in milligrams per deciliter (mg/dL). Normal range 61 to 199 mg/dL | 12 hours
  Differences in glucose (mg/dl) at the following time points, and also differences in the percentage of values within the normal range for each time point, for PBUF versus standard care.
  1. Final prime value (in the PBUF group after completion of PBUF and prior to cardio pulmonary bypass (CPB), in the control group prior to CPB)
  2. First measured levels on bypass - typically 10 minutes post initiation of bypass
  3. Last value on CPB
  4. Last value in OR
  5. First arrival to ICU
Sodium in milliequivalents per liter (mEq/L). Normal range 135 to 148 mEq/L | 12 hours
  Differences in sodium (mEq/L) at the following time points, and also differences in the percentage of values within the normal range for each time point, for PBUF versus standard care.
  1. Final prime value (in the PBUF group after completion of PBUF and prior to cardio pulmonary bypass (CPB), in the control group prior to CPB)
  2. First measured levels on bypass - typically 10 minutes post initiation of bypass
  3. Last value on CPB
  4. Last value in OR
  5. First arrival to ICU
Potassium in milliequivalents per liter (mEq/L). Normal range 3.2 to 4.5 mEg/L | 12 hours
  Differences in potassium (mEq/L) at the following time points, and also differences in the percentage of values within the normal range for each time point, for PBUF versus standard care.
  1. Final prime value (in the PBUF group after completion of PBUF and prior to cardio pulmonary bypass (CPB), in the control group prior to CPB)
  2. First measured levels on bypass - typically 10 minutes post initiation of bypass
  3. Last value on CPB
  4. Last value in OR
  5. First arrival to ICU
Lactate in milliequivalents per liter (mEq/L). Normal range 0.5 to 2.2 mEq/L | 12 hours
  Differences in lactate (mEq/L) at the following time points, and also differences in the percentage of values within the normal range for each time point, for PBUF versus standard care.
  1. Final prime value (in the PBUF group after completion of PBUF and prior to cardio pulmonary bypass (CPB), in the control group prior to CPB)
  2. First measured levels on bypass - typically 10 minutes post initiation of bypass
  3. Last value on CPB
  4. Last value in OR
  5. First arrival to ICU

SECONDARY OUTCOMES:
Osmolality in milli osmoles per kilogram (mOsm/Kg). Normal Range 276- 295 mOsm/kg | 12 hours
  Differences in osmolality in mOsm/Kg in final prime, first blood draw after CPB and on arrival to cardiac intensive care unit (CICU) for PBUF versus standard care.
Plasma free hemoglobin in milligrams per deciliter (mg/dL). Normal < 5 mg/dL. | 12 hours
  Differences in plasma free hemoglobin in mg/dL in final prime, first blood draw after CPB and on arrival to cardiac intensive care unit (CICU) for PBUF versus standard care.
Inotrope use | 72 hours
  Differences in vasoactive inotrope score between the PBUF and standard care groups at the following time points:
  i. Between cessation of CPB and admission to CICU as measured by vasoactive inotrope score (VIS) ii. In CICU as measure by VIS/ 24 hours for first 72 hours
Body wall edema as measured daily weights in kilograms (Kg) | Through study completion (until hospital discharge), an average of 15 days.
  Differences in body wall edema as measure by daily weights in Kg between the PBUF and standard care groups.
Body wall edema as measured daily weights in kilograms (Kg) | Through study completion (until hospital discharge) , an average of 15 days.
  Differences in body wall edema as measure by daily weights in Kg between the PBUF and standard care groups.
Initial ventilation duration in days and hours | Through study completion (until hospital discharge), an average of 15 days.
  Differences in ventilation duration, Initial (days, hours) until first extubation between the PBUF and standard care groups.
Reintubation as a proportion subjects needing reintubation in each group Reintubation | Through study completion (until hospital discharge), an average of 15 days.
  Difference in proportion of subjects requiring unplanned reintubation for respiratory failure between the PBUF and standard care groups.
Total ventilation duration (days, hours) | Through study completion (until hospital discharge), an average of 15 days.
  Difference in total ventilation duration (includes all periods on the ventilator including period following unplanned reintubation for respiratory failure between the PBUF and standard care groups.
Postoperative Cardiac intensive care unit (CICU) length of stay (LOS) in days, | Through study completion (until hospital discharge), an average of 15 days.
  Difference in postoperative CICU LOS in days between the PBUF and standard care groups.
Postoperative hospital LOS | Through study completion (until hospital discharge), an average of 15 days.
  Difference in postoperative hospital LOS in days between the PBUF and standard care groups.
Composite of major adverse events (Postoperative extra corporeal membrane oxygenation (ECMO), reoperation for bleeding, reoperation for low cardiac output state, circuit clotting events) and mortality. Yes or No | Through study completion (until hospital discharge), an average of 15 days.
  Difference in proportion subjects who have a composite event between the PBUF and standard care groups.

CONTACTS AND LOCATIONS:
Overall Officials: Meena Nathan, MD, MPH, Study Chair — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moore GL, Peck CC, Sohmer PR, Zuck TF. Some properties of blood stored in anticoagulant CPDA-1 solution. A brief summary. Transfusion. 1981 Mar-Apr;21(2):135-7. doi: 10.1046/j.1537-2995.1981.21281178147.x. PMID 7222197
- [Background] de Vroege R, Wildevuur WR, Muradin JA, Graves D, van Oeveren W. Washing of stored red blood cells by an autotransfusion device before transfusion. Vox Sang. 2007 Feb;92(2):130-5. doi: 10.1111/j.1423-0410.2006.00852.x. PMID 17298575
- [Background] Hall TL, Barnes A, Miller JR, Bethencourt DM, Nestor L. Neonatal mortality following transfusion of red cells with high plasma potassium levels. Transfusion. 1993 Jul;33(7):606-9. doi: 10.1046/j.1537-2995.1993.33793325059.x. PMID 8333025
- [Background] Baz EM, Kanazi GE, Mahfouz RA, Obeid MY. An unusual case of hyperkalaemia-induced cardiac arrest in a paediatric patient during transfusion of a 'fresh' 6-day-old blood unit. Transfus Med. 2002 Dec;12(6):383-6. doi: 10.1046/j.1365-3148.2002.00402.x. PMID 12473156
- [Background] O'Leary MF, Szklarski P, Klein TM, Young PP. Hemolysis of red blood cells after cell washing with different automated technologies: clinical implications in a neonatal cardiac surgery population. Transfusion. 2011 May;51(5):955-60. doi: 10.1111/j.1537-2995.2010.02935.x. Epub 2010 Nov 23. PMID 21091957
- [Background] Masalunga C, Cruz M, Porter B, Roseff S, Chui B, Mainali E. Increased hemolysis from saline pre-washing RBCs or centrifugal pumps in neonatal ECMO. J Perinatol. 2007 Jun;27(6):380-4. doi: 10.1038/sj.jp.7211748. Epub 2007 Apr 19. PMID 17443201
- [Background] Rao R, Georgieff MK. Iron in fetal and neonatal nutrition. Semin Fetal Neonatal Med. 2007 Feb;12(1):54-63. doi: 10.1016/j.siny.2006.10.007. Epub 2006 Dec 6. PMID 17157088
- [Background] Mumby S, Chaturvedi RR, Brierley J, Lincoln C, Petros A, Redington AN, Gutteridge JM. Iron overload in paediatrics undergoing cardiopulmonary bypass. Biochim Biophys Acta. 2000 Mar 17;1500(3):342-8. doi: 10.1016/s0925-4439(00)00003-x. PMID 10699376
- [Background] Jeffers A, Gladwin MT, Kim-Shapiro DB. Computation of plasma hemoglobin nitric oxide scavenging in hemolytic anemias. Free Radic Biol Med. 2006 Nov 15;41(10):1557-65. doi: 10.1016/j.freeradbiomed.2006.08.017. Epub 2006 Aug 25. PMID 17045924
- [Background] Vercaemst L. Hemolysis in cardiac surgery patients undergoing cardiopulmonary bypass: a review in search of a treatment algorithm. J Extra Corpor Technol. 2008 Dec;40(4):257-67. PMID 19192755
- [Background] Messent M, Sinclair DG, Quinlan GJ, Mumby SE, Gutteridge JM, Evans TW. Pulmonary vascular permeability after cardiopulmonary bypass and its relationship to oxidative stress. Crit Care Med. 1997 Mar;25(3):425-9. doi: 10.1097/00003246-199703000-00009. PMID 9118657
- [Background] Hackbarth RM, Eding D, Gianoli Smith C, Koch A, Sanfilippo DJ, Bunchman TE. Zero balance ultrafiltration (Z-BUF) in blood-primed CRRT circuits achieves electrolyte and acid-base homeostasis prior to patient connection. Pediatr Nephrol. 2005 Sep;20(9):1328-33. doi: 10.1007/s00467-005-1970-1. Epub 2005 Jun 10. PMID 15947984
- [Background] Delaney M, Axdorff-Dickey RL, Crockett GI, Falconer AL, Levario MJ, McMullan DM. Risk of extracorporeal life support circuit-related hyperkalemia is reduced by prebypass ultrafiltration. Pediatr Crit Care Med. 2013 Jul;14(6):e263-7. doi: 10.1097/PCC.0b013e31828a70c5. PMID 23823207
- [Background] Nagashima M, Imai Y, Seo K, Terada M, Aoki M, Shinoka T, Koide M. Effect of hemofiltrated whole blood pump priming on hemodynamics and respiratory function after the arterial switch operation in neonates. Ann Thorac Surg. 2000 Dec;70(6):1901-6. doi: 10.1016/s0003-4975(00)02024-5. PMID 11156092
- [Background] Grist G. Boiling the frog: the dangers of elevated sodium in blood primed pumps for infants. AmSECT Today.2012;Nov/Dec:5.
- [Background] Matte GS. Perfusion for Congenital Heart Surgery: Notes on Cardiopulmonary Bypass for a Complex Patient Population. Oxford: Wiley-Blackwell; 2015. Chapter 2, Page 27-32.